CLINICAL TRIAL: NCT02990650
Title: Outcomes Associated With Progressive Balance And Gait Training Using The KineAssist® Robot
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Shirley Ryan AbilityLab (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00001977
Record Dates: First submitted 2016-10-16; First posted 2016-12-13 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2016-10

CONDITIONS: Cerebrovascular Accident
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard physical therapist (Active Comparator): A combination of nine balance training tasks where the physical therapist provides guarding against loss of balance
  Interventions: Behavioral: Balance Task Training with therapist guarding support
- standard robotic guarding (Experimental): A combination of nine balance training tasks where the robotic system provides guarding against loss of balance
  Interventions: Behavioral: Balance task training with robotic guarding support
- challenge based robotic guarding (Experimental): A combination of nine balance training tasks where the robotic system provides guarding against loss of balance while the participant works at a level greater than their current balance capability
  Interventions: Behavioral: Challneged balance task training with robotic guarding support

INTERVENTIONS:
Behavioral: Balance Task Training with therapist guarding support — Nine balance tasks:
  1. long forward step
  2. forward reach
  3. push forward
  4. push backward
  5. step over hurdle
  6. step up on foam surface
  7. step up on solid surface
  8. sit-to-stand
  9. step onto slippery surface The therapist will provide guarding support
  Arms: Standard physical therapist
Behavioral: Balance task training with robotic guarding support — Nine balance tasks:
  1. long forward step
  2. forward reach
  3. push forward
  4. push backward
  5. step over hurdle
  6. step up on foam surface
  7. step up on solid surface
  8. sit-to-stand
  9. step onto slippery surface The guarding support will be provided by a robot
  Arms: standard robotic guarding
Behavioral: Challneged balance task training with robotic guarding support — Nine balance tasks where the subject is challenged to perform at a harder level of difficulty:
  1. long forward step
  2. forward reach
  3. push forward
  4. push backward
  5. step over hurdle
  6. step up on foam surface
  7. step up on solid surface
  8. sit-to-stand
  9. step onto slippery surface The guarding support will be provided by a robot
  Arms: challenge based robotic guarding

SUMMARY:
Using a randomized controlled research design, compare walking outcomes resulting from gait and balance training with standard physical therapist interaction versus training with the addition of a KineAssist® robotic system that provides for safety and freedom of movement.

DETAILED DESCRIPTION:
Several studies have investigated the use of balance and gait training and have demonstrated significant improvements in walking speed with trained stroke survivors. The inherent risks associated with balance and gait training requires the therapist to be vigilant with providing safety and support during challenging tasks. As a result, consumers are not challenged to their furthest limits and therapists put an inordinate amount of physical effort into safety control. KineAssist® Design, LLC in collaboration with Rehabilitation Institute of Chicago, developed the KineAssist® Balance and Gait Training System (KineAssist®). The KineAssist® is a novel device that allows full freedom of motion for the trunk and pelvis during gait and balance tasks, with additional postural control to enhance balance stability. These functions are available while the device follows the individual overground with minimal interference. The availability of postural control during complex and omnidirectional movement tasks allows the clinician to guarantee consumer safety and body weight support while at the same time provide graded task challenges to the fullest limits of the consumers capabilities. This KineAssist® is revolutionary in that it is the first device that is fully interactive and responsive to the movements and intentions of both the consumer and the therapist during overground challenging balance and gait activities.

Accordingly, the long-term objective of this research is to test the efficacy of robotically enhanced, progressive gait and balance training for improving walking outcomes post-stroke. The following two aims are designed to test whether the KineAssist® provides a more challenging training environment than is typical with physical therapy, and then compares walking outcomes as a result of long-term (6 weeks) training.

Aim: Using a randomized controlled research design, compare walking outcomes resulting from gait and balance training with standard physical therapist interaction versus training with the addition of a KineAssist®t.

Overall, these studies are an important advance for the development of effective clinical interventions for individuals with impaired locomotor ability post-stroke. This study will provide critical information on physiological effects and clinical outcomes and provide important evidence for the use of this new class of robotic technology that accommodates both the clinician and the consumer in stroke rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* > 6 months post-stroke
* post-stroke hemiparesis
* 1.0 m/sec or slower walking speed

Exclusion Criteria:

* musculoskeletal injury
* recent history of cardiac event
* other neurological disease or disorders
* inability to follow three-step commands
* uncontrolled diabetes and/or high blood pressure

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-10; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Mean time of 10 meter walk test at baseline | baseline
Mean time of 10 meter walk test at 3 weeks post baseline | 3 weeks post baseline
Mean time of 10 meter walk test at 6 weeks at end of training | 6 weeks post baseline
Mean time of 10 meter walk test at 6 months post training | 6 months post end of training
Mean time of 6 minute walk test at baseline | baseline
Mean time of 6 minute walk test at 3 weeks post baseline | 3 weeks post baseline
Mean time of 6 minute walk test at 6 weeks post baseline (end of training) | 6 weeks post baseline (end of training)
Mean time of 6 minute walk test at 6 months post training | 6 months post end of training (7.5 months post baseline)
Mean Berg Balance Scale score at baseline | baseline
  The Berg Balance Scale has a range of 56 (best) to 14 (worst). There are 14 different balance tasks each with a an assigned rank of 1 - 4 (1, 2, 3, 4). 1 is the worst performance and 4 is the best.
Mean Berg Balance Scale score at 3 weeks post baseline | 3 weeks post baseline
  The Berg Balance Scale has a range of 56 (best) to 14 (worst). There are 14 different balance tasks each with a an assigned rank of 1 - 4 (1, 2, 3, 4). 1 is the worst performance and 4 is the best.
Mean Berg Balance Scale score at 6 weeks post baseline (end of training) | 6 weeks post baseline
  The Berg Balance Scale has a range of 56 (best) to 14 (worst). There are 14 different balance tasks each with a an assigned rank of 1 - 4 (1, 2, 3, 4). 1 is the worst performance and 4 is the best.
Mean Berg Balance Scale score at 6 months post end of training | 6 months post end of training (7.5 months post baseline)
  The Berg Balance Scale has a range of 56 (best) to 14 (worst). There are 14 different balance tasks each with a an assigned rank of 1 - 4 (1, 2, 3, 4). 1 is the worst performance and 4 is the best.

CONTACTS AND LOCATIONS:
Locations (1):
- Locomotor Control Lab, Birmingham, Alabama, United States